CLINICAL TRIAL: NCT03490500
Title: Improving the Headache Management Care in the Emergency Unit by Using a Biological Marker: S100B Protein.
Brief Title: Using the S100B Protein for Emergency Headache Management Care (S100)
Acronym: S100
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-CHITS-07; 2018-A00070-55 (Other: Id-RCB)
Record Dates: First submitted 2018-03-26; First posted 2018-04-06 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Headache, Migraine; Hemorrhage
Keywords: protein S100B; negative predictive value; headache; intracranial hemorrhage
MeSH Terms: conditions — Migraine Disorders; Hemorrhage; Headache; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample for protein S100B dosage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- S100B protein dosage: Biological

SUMMARY:
The purpose of this study is to determine the negative predictive value of protein S100B that could exclude subarachnoid and intracranial haemorrhage for patient that present severe headache within the last 3 hours.

DETAILED DESCRIPTION:
This study will be proposed to every patient that correspond to eligibility criteria, such as presenting a severe headache (Visual Analog Scale ≥ 6/10) within 3 hours before arriving to the emergency.

After signing the informed consent, a blood sample will be taken in order to dosage S100B protein of each patient, and then they will have a brain scan.

The trial ends after the brain scan for each patient. Results of brain scans will be compared with results of S100B dosage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years-old
* Patient presenting at the Emergency Service a non-traumatic severe headache lasting for less than 3 hours. The severity is defined as a VAS ≥ 6/10
* Blood sample can be taken within 1 hour following the emergency admission
* VAS > 6 or Glasgow < 8
* Signed and dated informed consent by patient, or trusted person, or family

Exclusion Criteria:

* Patient presenting headache after head trauma
* Pregnant or breastfeeding women
* Patient with a pathology causing the elevation of PS100B's rate such as Alzheimer's disease, Creuzfeld-Jacob's disease, Multiple Sclerosis, cerebral tumour, trisomy 21, melanoma (diabetes excluded)
* Patient covered by social security regimen or equivalent
* Patient under guardianship (legal protection)
* Patient deprived of liberty by court or administrative order
* Any condition that could influence PS100B's dosage results according to the physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be recruited in the emergency unit
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Evaluate the interest of PS100B dosage in the severe headache therapeutic management | 15 months
  Negative predictive value of PS100B dosage below the reference value of 0.10 µG/L for intracerebral haemorrhage lesion

SECONDARY OUTCOMES:
Frequency of Intracranial Bleeding in patient with severe headache | 15 months
  Incidence of intracranial bleeding in patient with severe headache
Frequency of subarachnoid hemorrhage in patient with severe headache | 15 months
  Incidence of subarachnoid haemorrhage in patient with severe headache
Frequency of intracranial haemorrhage in migraine patient with severe headache at inclusion | 15 months
  Incidence of intracranial haemorrhage in migraine patient with severe headache at inclusion
Evaluate the number of lumbar puncture that could have been avoided | 15 months
  The ratio of patient with a normal scan and a PS100 dosage < 0.10µg/L, on patient eligible for lumbar puncture according to the usual practice
Evaluate the number of cerebral scan that could have been avoided | 15 months
  The ratio of patient with a normal scan and a PS100 dosage < 0.10 µg/L, on patient eligible for cerebral scan according to the usual practice
Evaluate the number of lumbar puncture's complications that could have been avoided. | 15 months
  The ratio of patients with PS100 < 0.10µg/L and normal cerebral scan on the total number of patients included

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Renard, MD, Study Director — Hôpital d'instruction des armées Sainte-Anne
Locations (3):
- France (3):
  - Hôpital d'Instruction des Armées Laveran, Marseille, Bouches-du-Rhône
  - Hôpital d'Instruction des Armées Sainte Anne, Toulon, Var
  - Centre Hospitalier Intercommunal de Toulon La Seyne-sur-Mer, Toulon, Var

IPD SHARING:
Plan to Share IPD: No
There is no IPD sharing plan

REFERENCES:
- [Background] Latinovic R, Gulliford M, Ridsdale L. Headache and migraine in primary care: consultation, prescription, and referral rates in a large population. J Neurol Neurosurg Psychiatry. 2006 Mar;77(3):385-7. doi: 10.1136/jnnp.2005.073221. PMID 16484650
- [Background] Edlow JA, Panagos PD, Godwin SA, Thomas TL, Decker WW; American College of Emergency Physicians. Clinical policy: critical issues in the evaluation and management of adult patients presenting to the emergency department with acute headache. Ann Emerg Med. 2008 Oct;52(4):407-36. doi: 10.1016/j.annemergmed.2008.07.001. PMID 18809105
- [Background] Biberthaler P, Linsenmeier U, Pfeifer KJ, Kroetz M, Mussack T, Kanz KG, Hoecherl EF, Jonas F, Marzi I, Leucht P, Jochum M, Mutschler W. Serum S-100B concentration provides additional information fot the indication of computed tomography in patients after minor head injury: a prospective multicenter study. Shock. 2006 May;25(5):446-53. doi: 10.1097/01.shk.0000209534.61058.35. PMID 16680008
- [Background] Gilbert JW, Johnson KM, Larkin GL, Moore CL. Atraumatic headache in US emergency departments: recent trends in CT/MRI utilisation and factors associated with severe intracranial pathology. Emerg Med J. 2012 Jul;29(7):576-81. doi: 10.1136/emermed-2011-200088. Epub 2011 Aug 19. PMID 21856709
- [Background] Morgenstern LB, Huber JC, Luna-Gonzales H, Saldin KR, Grotta JC, Shaw SG, Knudson L, Frankowski RF. Headache in the emergency department. Headache. 2001 Jun;41(6):537-41. doi: 10.1046/j.1526-4610.2001.041006537.x. PMID 11437887
- [Background] Edlow JA, Caplan LR. Avoiding pitfalls in the diagnosis of subarachnoid hemorrhage. N Engl J Med. 2000 Jan 6;342(1):29-36. doi: 10.1056/NEJM200001063420106. No abstract available. PMID 10620647
- [Result] Muller P, Mitri F, Houlle A, Vidal PO, Gasperini G, Cazes N, Renard A. S100ss protein for non-traumatic subarachnoid hemorrhage diagnosis. Am J Emerg Med. 2022 Jul;57:39-41. doi: 10.1016/j.ajem.2022.04.030. Epub 2022 Apr 25. PMID 35500528